CLINICAL TRIAL: NCT05848531
Title: Advantage of Clonidine With Morphine In Patient Controlled Analgesia Pump for the Treatment of Vaso-occlusive Crisis in Sickle Cell Disease Patients
Brief Title: Clonidine With Morphine in Patient Controlled Analgesia Pump in Vaso-Occlusive Crisis in Sickle Cell Disease Patient
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Lara Chow Yuen, Principal Investigator, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B0762023230104
Record Dates: First submitted 2023-03-30; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episode in Sickle Cell Disease
Keywords: Clonidine; Morphine; Acute Pain management; patient controlled analgesia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Double Blinded, randomised, prospective
Who Masked: Participant, Care Provider, Investigator
Masking Description: Unmarked bags of products, randomised before administration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine (No Intervention): Standard Morphine PCIA
- Clonidine and Morphine (Experimental): Morphine Associated with Clonidine PCIA
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — Comparing Clonidine with Morphine PCIA for the treatment of Vaso-Occlusive crisis in Sickle Cell disease patient
  Other Names: Catapressan
  Arms: Clonidine and Morphine

SUMMARY:
Vaso-occlusive crisis are highly painful in Sickle-cell patients. Morphine is the treatment of choice for this pain. Various adjuncts have been studied for the treatment of vaso-occlusive crisis.

The investigators aimed to study the effect of clonidine associated with morphine in PCIA (patient controlled intravenous analgesia pumps) regimen. The investigators will compare it to the morphine alone in PCIA for the treatment of vaso-occlusive pain.

The investigators will measure the morphine consumption of all patient, the impact on the apparition of the morphine secondary effect and on inflammation biomarkers and the biopsychosocial respond.

Each patient will be hospitalized and follow by haematologist from the hospital, pain doctors and nurses.

It will be a double blind randomised, prospective study. The randomisation will be done by the pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Vaso-Occlusive Crisis In Sickle Cell disease Patients

Exclusion Criteria:

* Minor
* Patient's refusal
* Pregnancy
* Contr-indication Clonidine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Morphine Consumption | Up to two weeks
  Morphine Consumption during hospitalisation

SECONDARY OUTCOMES:
Numerical Rating Scale | Up to two weeks
  Pain Score scale from 0 to ten during and after treatment
Biology markers | Up to two weeks
  Inflammatory biology markers (CRP,IL-6) and Hemolysis (LDH)
Biopsychosocial model / ASCQ-ME questionary | Up to two weeks
  Evaluation of the biopsychosocial model. There are seven different themes of 4 to 7 questions each (pain intensity, pain episodes, sleep impact, social impact, emotional impact, medical history and stiffness)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Saint-Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kenney MO, Smith WR. Moving Toward a Multimodal Analgesic Regimen for Acute Sickle Cell Pain with Non-Opioid Analgesic Adjuncts: A Narrative Review. J Pain Res. 2022 Mar 31;15:879-894. doi: 10.2147/JPR.S343069. eCollection 2022. PMID 35386424